CLINICAL TRIAL: NCT04544774
Title: The Role of the Nasal Allergen Provocation Test in Starting and Monitoring Allergen Immunotherapy: An Academic Multicentre Clinical Study
Brief Title: The Role of the Nasal Allergen Provocation Test in Starting and Monitoring Allergen Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, prof. dr. Laura Van Gerven, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s63711
Record Dates: First submitted 2020-08-19; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Perennial Allergic Rhinitis; Seasonal Allergic Rhinitis; Local Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergic rhinitis patients: Patients with persistent or intermittent allergic rhinitis complaints, confirmed by skin prick tests and/or immunocap for specific IgEs, that start with AIT treatment.
  Interventions: Drug: AIT; Diagnostic Test: NAPT

INTERVENTIONS:
Drug: AIT — AIT for airborn allergens (SCIT/SLIT)
Diagnostic Test: NAPT — NAPT test with airborn allergens ( HDM, Threes, Grasses)

SUMMARY:
This prospective multicentric academic NAPT study aims to compile a database of all patients who initiate immunotherapy.

The NAPT will take place before, during and after AIT to evaluate the cost and effectiveness of the treatment. The study consists of 4 visits and 2 telephone contacts that are repeated annually for 3 years.

This study will be conducted in 2 hospitals: UZ Leuven and AZ ST. Jan Brugge on the consultation Ear, Nose and Throat Diseases (ENT) and the department of Internal Medicine / Allergology

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and ≤60 years
* Persistent or intermittent allergic rhinitis complaints, confirmed by SPT and/of immunocap for the specific IgEs.

OR suspected local allergic rhinitis

* Patients who start with AIT treatment
* The patient must be motivated and willing to come to all visits
* The patient must be able to understand and sign the informed consent

Exclusion Criteria:

* Uncontrolled asthma
* Conditions affecting the functioning of the immune system (eg: immune deficiencies, malignancies, autoimmune diseases)
* Use of β-blockers, immunosuppressants or ACE inhibitors
* Hypersensitivity to aluminum hydroxide and/or hypersensitivity to any of the excipients in AIT
* Anaphylaxis after allergen challenge in the past
* Acute rhinosinusitis in the last 12 weeks
* Recent surgery on the nose and/or paranasal sinuses in the last 12 weeks
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with persistent and intermittent allergic rhinitis who start with AIT treatment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of AIT treatment assessed by the change in the blood concentration in total en specific IgE . | before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing blood results, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the Lebelscore. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing the Lebelscores ,assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  Lebelscore has a range between 0 and 12.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the SNOT-22. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing SNOT-22, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  SNOT-22 is sino-nasal outcome test with 22 items which ranges from 0 to 110.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the VAS. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing VAS, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  The visual analogue scale (VAS) ranges from 0 to 10cm for every item.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the TNSS. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing TNSS, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  Total nasal symptom score (TNSS) ranges from 0 to 12.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the ACT. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing ACT, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  ACT is the Asthma control test with scores between 0 and 25. The higher the score the better.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the RQLQ. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing RQLQ, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  RQLQ is the rhinoconjunctivits quality of life questionnaire with scores between 0 and 168.
  The higher the score of these questionnaires the more discomfort.
The effectiveness of AIT treatment assessed by the change in quality of life meassured by the TRE. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing TRE, assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up).
  TRE is the therapeutic response evaluation and will be scored between 'much better' and 'much worse'.
The effectiveness of AIT treatment assessed by the change in the PNIF value. | Before start AIT, every 6 months en after 3 years
  The effectiveness of AIT treatment will be analysed by comparing PNIF values assessed by the NAPT tests, before, during (every 6 months after starting AIT) and after end of treatment (approximately 3 years after start-up). PNIF is the peak nasal inspiratory flow with a value between 0 and 370 l/min). The higher the value the less congested the nose is.

SECONDARY OUTCOMES:
Calculating the cost savings by desensitizing poly-sensitized patients only to the allergen to which they respond most strongly in the NAPT test. | 3 years
Calculating the cost savings by timely stopping AIT treatment in non-responders, which we can define as patients who do not experience subjective or objective improvement after 1 year of treatment. | 3 year

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven, Vlaam Brabant
  - AZ Sint-Jan, Bruges

IPD SHARING:
Plan to Share IPD: No